CLINICAL TRIAL: NCT00649025
Title: A Randomized, Double-blind, Active-controlled, Parallel Group, Stratified, Multi-center, 12-Week Study Comparing the Safety and Efficacy of Fluticasone and Formoterol Combination (FlutiForm™ 250/10ug Twice Daily) in a Single Inhaler (SkyePharma HFA pMDI) With the Administration of Fluticasone (250ug Twice Daily) Alone in SkyePharma HFA pMDI and Flovent® HFA pMDI in Adolescent and Adult Patients With Moderate to Severe Asthma
Brief Title: A Study Comparing the Safety and Efficacy of Fluticasone and Formoterol Combination (FlutiForm™) With Fluticasone or Flovent to Treat Moderate to Severe Asthma in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Collaborators: Abbott (Industry); MDS Pharma Services (Industry)
Responsible Party: SkyePharma AG, SkyePharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKY2028-3-005
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Asthma
Keywords: Asthma; Asthma Moderate to Severe
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): FlutiForm 250/10ug
  Interventions: Drug: FlutiForm 250/10
- 2 (Active Comparator): SKP Fluticasone 250ug
  Interventions: Drug: SKP-Fluticasone
- 3 (Active Comparator): Flovent Fluticasone HFA
  Interventions: Drug: Flovent Fluticasone HFA

INTERVENTIONS:
Drug: FlutiForm 250/10 — SKP FlutiForm 250/10ug is a HFA pMDI that delivers 125ug of Fluticasone propionate per actuation and 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Arms: 1
Drug: SKP-Fluticasone — SKP Fluticasone 250 ug is a HFA pMDI that delivers 125ug of Fluticasone propionate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Arms: 2
Drug: Flovent Fluticasone HFA — Flovent 250 ug HFA is a pMDI that delivers after priming 125ug of Fluticasone propionate per actuation. Patients will take 2 actuations BID for 12 weeks.
  Other Names: Flovent
  Arms: 3

SUMMARY:
The medications being used in this study are individually approved by the Food and Drug Administration (FDA). The medication under investigation is a combination of two medications in one inhaler. The purpose of this study is to determine how well your asthma is controlled when taking one of the three treatment.

DETAILED DESCRIPTION:
This Phase 3 randomized, double-blind, active-controlled, parallel group, stratified, multi-center study will evaluate the safety and efficacy of FlutiForm (250/10ug) after twice daily dosing over 12 weeks delivered by SKP HFA pMDI compared with Fluticasone propionate (250ug of twice daily) delivered by SKP HFA pMDI and Flovent® Fluticasone 250ug HFA pMDI in adolescent and adult patients with moderate to severe asthma. Only steroid-requiring patients (inhaled steroid regimen stable for at least 4 weeks prior to the Screening Visit at a dose not greater than 500ug/day Fluticasone propionate or equivalent) will be eligible. All patients will undergo a Run-In Period of 14 ± 3 days during which they will receive asthma maintenance therapy using Fluticasone HFA pMDI (Flovent® HFA 50 ug/actuation: 100µg/day (one inhalation twice daily) if they were using less than or equal to 250mg/day Fluticasone propionate or equivalent inhaled steroid, or 200ug/day (two inhalations twice daily) if they were using greater than 250ug/day Fluticasone propionate or equivalent inhaled steroid prior to the Screening Visit.). The use of rescue Salbutamol (Albuterol) pMDI will be permitted for all patients as needed for the control of worsening asthma symptoms during the Run-In Period. At the Baseline Visit (Week 0) following the Run-In period, eligible patients will be randomized to the treatment groups. Treatment assignment will be stratified according to their Baseline FEV1 % predicted (40-60% or >60-80%).Study drug will be administered twice daily over a 12-week period. Patient visits will occur at Weeks 2, 4, 8, and 12 during which assessments (including serial PFTs up to 4 hours) will be made. In a subset of at least 66 patients (22 patients per treatment group) from selected centers, post-dose 12-hour serial PFTs will be performed at Baseline, Weeks 2 and 12. During the Treatment Period, patients may only take their blinded study medication; all other asthma medications will be withheld for the duration of the Treatment Period. However, the use of rescue Salbutamol (Albuterol) pMDI will be permitted in all patients as needed during the Treatment Period for the control of worsening asthma symptoms.

ELIGIBILITY:
Main Inclusion Criteria:

* ≥ Age 12 years at the Screening Visit.
* History of asthma for 12 months prior to the Screening Visit.
* Documented use of an inhaled corticosteroid for at least 4 weeks prior to the Screening Visit.
* Steroid-requiring patient
* patients must demonstrate (1) an FEV1 of 40% to 80% (inclusive) of predicted normal values at both the Screening and Baseline Visits and (2) documented reversibility within 12 months of the Screening Visit, defined as a ≥ 15%

Main Exclusion Criteria:

* Life-threatening asthma within the past year or during the Run-In Period.
* History of systemic (oral or injectable) corticosteroid medication within 3 months before the Screening Visit.
* An upper or lower respiratory infection within 4 weeks prior to the Screening Visit or during the Run-In Period.
* Significant, non-reversible, pulmonary disease (e.g., chronic obstructive pulmonary disease [COPD], cystic fibrosis, bronchiectasis).
* A smoking history equivalent to "10 pack years" (i.e., at least 1 pack of 20 cigarettes /day for 10 years or 10 packs/day for 1 year, etc.).
* Current smoking history within 12 months prior to the Screening Visit.
* Previous exposure to FlutiForm

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy in terms of the Formoterol fumarate component of SKP FlutiForm HFA pMDI (250/10ug) compared to SKP Fluticasone HFA pMDI (250ug), on the change in FEV1 from morning pre-dose at Baseline (Week 0) to 2 hours post-dose at Week 12. | Week 0 and 12 visits

SECONDARY OUTCOMES:
Demonstrate the efficacy of SKP FLUTIFORM HFA pMDI (250/10ug) compared to FLOVENT® Fluticasone pMDI (250ug) on the change in FEV1 from morning pre-dose at Baseline (Week 0) to 2 hours post-dose at Week 12. | Week 0 and 12 visits
Demonstrate the efficacy of SKP FLUTIFORM HFA pMDI (250/10ug) using other pulmonary function tests (PFTs), and clinical endpoints. | Whole duration of study
Assess the safety profile of SKP FLUTIFORM HFA pMDI (250/10ug twice daily) using incidence of adverse events, and changes in electrocardiograms, clinical laboratory tests and vital signs. | Whole duration of study
To assess the 12-hour serial FEV1 area under the curve (AUC) in a subset population (in a minimum of 66 patients). | Week 0; 2 and 12 visits

CONTACTS AND LOCATIONS:
Locations (72):
- United States (21):
  - Investigational site, Scottsdale, Arizona
  - Investigational Site, Tempe, Arizona
  - Investigational Site, Encinitas, California
  - Investigational site, Long Beach, California
  - Investigational site, Orange, California
  - Investigational Site, Oldsmar, Florida
  - Investigational Site, Indianapolis, Indiana
  - Investigational site, Crestview Hills, Kentucky
  - Investigational Site, Metarie, Louisiana
  - Investigational site, North Dartmouth, Massachusetts
  - Investigational Site, Wellesley Hills, Massachusetts
  - Investigational site, Elizabeth City, North Carolina
  - Investigational Site, Akron, Ohio
  - Investigational site, Cincinnati, Ohio
  - Investigational Site, Portland, Oregon
  - Investigational Site, East Providence, Rhode Island
  - Investigational site, Providence, Rhode Island
  - Investigational Site, Austin, Texas
  - Investigational site, El Paso, Texas
  - Investigational site, Richmond, Virginia
  - Investigational Site, West Allis, Wisconsin
- Argentina (7):
  - Investigational Site, Bahía Blanca
  - Investigational Site, Buenos Aires
  - Investigational Site, Caba
  - Investigational Site, Provincia de Buenos Aires
  - Investigational Site, Salta
  - Investigational Site, San Miguel de Tucumán
  - Investigational Site, Santa Fe
- Chile (3):
  - Investigational Site, Concepción
  - Investigational Site, Rancagua
  - Investigational Site, Santiago
- Hungary (4):
  - Investigational Site, Budapest
  - Investigational Site, Deszk
  - Investigational Site, Miskolc
  - Investigational Site, Pécs
- Mexico (10):
  - Investigational Site, Chihuahua City
  - Investigational Site, Guerrero
  - Investigational Site, Jalisco
  - Investigational Site, Luis Encinas S/N
  - Investigational Site, Mexico City
  - Investigational Site, Michoacán
  - Investigational Site, Nuevo León
  - Investigational Site, Puebla City
  - Investigational Site, San Bernardino
  - Investigational Site, Tabasco
- Peru (4):
  - Investigational Site, Cusco
  - Investigational Site, Jesus Maria
  - Investigational Site, Lima
  - Investigational Site, Lima Cercado
- Poland (5):
  - Investigational Site, Gdansk
  - Investigational Site, Krakow
  - Investigational Site, Lodz
  - Investigational Site, Rzeszów
  - Investigational Site, Wroclaw
- Romania (5):
  - Investigational Site, Brasov
  - Investigational Site, Bucharest
  - Investigational Site, Craiova
  - Investigational Site, Palazu Mare
  - Investigational Site, Timișoara
- South Africa (6):
  - Investigational Site, Bloemfontein
  - Investigational Site, Cape Town
  - Investigational Site, Durban
  - Investigational Site, Pretoria
  - Investigational Site, Somerset West
  - Investigational Site, Tygerberg
- Ukraine (7):
  - Investigational Site, Dnipropetrovsk
  - Investigational Site, Donetsk
  - Investigational Site, Kharkiv
  - Investigational Site, Kiev
  - Investigational Site, Lviv
  - Investigational Site, Vinnytsia
  - Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Pertseva T, Dissanayake S, Kaiser K. Superiority of fluticasone propionate/formoterol fumarate versus fluticasone propionate alone in patients with moderate-to-severe asthma: a randomised controlled trial. Curr Med Res Opin. 2013 Oct;29(10):1357-69. doi: 10.1185/03007995.2013.825592. Epub 2013 Aug 20. PMID 23865726